CLINICAL TRIAL: NCT04538716
Title: Orbital Fat Graft Retroseptal Transconjunctival Blepharoplasty for Treatment of Groove in the Infraorbital Region
Brief Title: Retroseptal Transconjunctival Blepharoplasty for GIR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Benha University (Other)
Responsible Party: Principal Investigator, Tarek Roshdy mohamed Mahgoub ELhamaky, lecturer, Benha University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Hamaky6
Record Dates: First submitted 2020-08-31; First posted 2020-09-04 (Actual); Last update posted 2023-11-15 (Actual); Status verified 2023-11

CONDITIONS: Eyelid Diseases
Keywords: tear trough, blepharoplasty,orbital fat
MeSH Terms: conditions — Eyelid Diseases

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SVF-gel (Experimental): Transconjunctival blepharoplasty associated with associated with stromal vascular fraction gel (SVF-gel)
  Interventions: Procedure: transconjunctival lower blepharoplasty
- fat transposition (Experimental): Transconjunctival blepharoplasty associated with fat transposition
  Interventions: Procedure: transconjunctival lower blepharoplasty

INTERVENTIONS:
Procedure: transconjunctival lower blepharoplasty — transconjunctival lower blepharoplasty associated with stromal vascular fraction gel (SVF-gel)

SUMMARY:
The tear trough deformity is a challenging cosmetic condition.surgical treatment and filling are good treatment options

DETAILED DESCRIPTION:
Procedure is lower eyelid transconjunctival Blepharoplasty associated with stromal vascular fraction gel (SVF-gel) or fat transposition

ELIGIBILITY:
Inclusion Criteria:

* tear trough deformity

Exclusion Criteria:

* Eyelid diseases and previous eyelid surgery

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2019-08-01 (Actual); Primary Completion 2023-11-01 (Actual); Study Completion 2023-11-10 (Actual)

PRIMARY OUTCOMES:
skin-periosteal depth | 2 years
  measure skin-periosteal depth

SECONDARY OUTCOMES:
global aesthetic improvement scale | 2 years
  calculate scale score from score 1 (exceptional improvement) to score 5 (worsening patient)

CONTACTS AND LOCATIONS:
Overall Officials: TAREK ELHAMAKY, MD, Principal Investigator — Benha university faculty of medicine
Locations (1):
- INMC, Abu Dhabi, United Arab Emirates

REFERENCES:
- [Derived] Elhamaky TR. Orbital fat graft retroseptal transconjunctival blepharoplasty for treatment of groove in the infraorbital region. Int Ophthalmol. 2024 May 6;44(1):217. doi: 10.1007/s10792-024-03148-z. PMID 38705907